CLINICAL TRIAL: NCT02725138
Title: The Efficacy of Lactobacillus Acidophilus and Lactobacillus Rhamnosus in the Modification of Gut Microbiota and Reduction of Helicobacter Pylori Bacterial Load- a Double Blind, Placebo Controlled, Randomized Trial
Brief Title: Efficacy of Probiotics in the Gut Microbiota and H Pylori Density
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Statistical Center, NTUHCTC (Other)
Collaborators: Taiwan Sugar Cooperation Company (Unknown)
Responsible Party: Sponsor-Investigator, Statistical Center, NTUHCTC, Attending physician, National Taiwan University Hospital
Organization: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201511071RIPA
Record Dates: First submitted 2016-03-27; First posted 2016-03-31 (Estimated); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Helicobacter
Keywords: Helicobacter pylori; probiotic; bacterial density
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Experimental): subjects will be treated with probiotic containing Lactobacillus acidophilus，Lactobacillus rhamnosus, 1pack, twice daily, for 4 weeks
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): subjects will be treated with placebo without Lactobacillus acidophilus，Lactobacillus rhamnosus, 1pack, twice daily, for 4 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotic containing Lactobacillus acidophilus and Lactobacillus rhamnosus produced by the Taiwan Sugar Cooperation, 1pack, twice daily, for 4 weeks
  Arms: Probiotic
Other: Placebo — Placebo without Lactobacillus acidophilus and Lactobacillus rhamnosus produced by the Taiwan Sugar Cooperation, 1pack, twice daily, for 4 weeks
  Arms: Placebo

SUMMARY:
We aimed to assess the efficacy of Lactobacillus acidophilus and Lactobacillus rhamnosus in the reduction of bacterial load of H. pylori and in the modification of gut microbiotia in this double blind, placebo controlled, randomized trial.

DETAILED DESCRIPTION:
Subjects: Adult subjects aged 20 or greater with moderate to high bacterial load of H. pylori defined as a DOB value greater than 10 will be eligible to this trial. We will screen 150 subjects and it is estimated that 40 H. pylori infected subjects will be eligible. Eligible subjects will be randomized to receive probiotic (Lactobacillus acidophilus and Lactobacillus rhamnosus) or placebo, one pack twice daily, for 28 days. The primary outcome was the reduction in H. pylori load of greater than 20% than baseline. The secondary outcome was the impact of the probiotic on the gut microbiota and the adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects aged 20 or greater with moderate to high bacterial load of H. pylori defined as a DOB value greater than 10 will be eligible to this trial

Exclusion Criteria:

* history of gastrectomy and colectomy
* severe underlying illness, such as malignancy, ESRD, liver failure, etc
* allergy to probiotics
* symptomatic patients who need PPI, antibiotics, or other probiotics
* pregnancy and lactating women
* unable to cooperate with the protocol

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Reduction of bacterial load of H. pylori | after 4 weeks of treatment

SECONDARY OUTCOMES:
changes in gut microbiota | after 4 weeks of treatment
adverse effects | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Ming Liou, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen MJ, Chen CC, Huang YC, Tseng CC, Hsu JT, Lin YF, Fang YJ, Wu MS, Liou JM; Taiwan Gastrointestinal Disease, Helicobacter Consortium. The efficacy of Lactobacillus acidophilus and rhamnosus in the reduction of bacterial load of Helicobacter pylori and modification of gut microbiota-a double-blind, placebo-controlled, randomized trial. Helicobacter. 2021 Dec;26(6):e12857. doi: 10.1111/hel.12857. Epub 2021 Oct 27. PMID 34708471